CLINICAL TRIAL: NCT06849856
Title: Clinical and Biochemical Evaluation of the Efficacy of Different Non-Surgical Peri-implantitis Treatment Approaches
Brief Title: Evaluation of the Efficacy of Different Non-Surgical Peri-implantitis Treatment Approaches
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Meltem Ozdemir Kabalak, Instructor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THD-2023-20873
Record Dates: First submitted 2025-01-20; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-02

CONDITIONS: Periimplantitis
Keywords: peri-implantitis, airflow
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment of peri-implantitis using titanium curette (Active Comparator): Non-surgical peri-implantitis treatment will be performed using titanium curettes suitable for use on implant surfaces
  Interventions: Procedure: non-surgical peri-implantitis therapy with titanium curette
- Treatment of peri-implantitis using Airflow device (Experimental): Non-surgical peri-implantitis treatment will be performed using erythritol powder with Airflow device
  Interventions: Device: non-surgical peri-implantitis therapy with airflow device
- Treatment of peri-implantitis using titanium curette + Airflow device (Experimental): Non-surgical peri-implantitis treatment will be performed using titanium curette and erythritol powder with Airflow device
  Interventions: Device: non-surgical peri-implantitis therapy with airflow device; Procedure: non-surgical peri-implantitis therapy with titanium curette

INTERVENTIONS:
Device: non-surgical peri-implantitis therapy with airflow device — Airflow device with erythritol powder will be used in the treatment of non-surgical peri-implantitis
  Arms: Treatment of peri-implantitis using Airflow device; Treatment of peri-implantitis using titanium curette + Airflow device
Procedure: non-surgical peri-implantitis therapy with titanium curette — Titanium curette will be used for non-surgical treatment of peri-implantitis
  Arms: Treatment of peri-implantitis using titanium curette; Treatment of peri-implantitis using titanium curette + Airflow device

SUMMARY:
Peri-implant diseases, which are the most common biological complications of dental implants, are inflammatory diseases characterized by soft tissue inflammation and loss of supporting bone tissue in the tissues around the implant. The most basic factor in the onset of peri-implant diseases is bacterial biofilm formation. Therefore, the gold standard in its treatment is plaque removal. It has been stated that mechanical treatments with conventional plaque removal methods, usually applied using curettes in the treatment of peri-implantitis, are unpredictable and that positive clinical results are valid for short periods such as 6-12 months. This result can be explained by the inability to provide sufficient debridement on the rough implant surface. For this reason, it has been shown that the use of air abrasion systems based on the principle of cleaning the surfaces by applying an abrasive powder with compressed air may be beneficial in order to increase the success of the treatment. When the literature is reviewed, it is seen that there is no standard clinical protocol for the use of air abrasion devices as a mechanical debridement method for non-surgical peri-implantitis treatment. In the pathogenesis of peri-implant disease, cytokines that manage the inflammatory process play a major role. RANK ligand (RANKL), osteoprotegerin (OPG) and TWEAK are biomarkers that play a role in bone metabolism. Examination of cytokines and such biomarkers that play a role in bone metabolism in the peri-implant crevicular fluid (PIOS) at the initial stage and during the post-treatment follow-up processes and recording clinical findings may be useful in evaluating the effects of alternative treatment methods on disease control. For this purpose, it is planned to include 60 patients aged between 18-65 with dental implants with a probing depth of 6 mm or more in one or more areas of the mouth in the study. Patients will be randomized into 3 groups as A: Non-surgcal treatment with titanium curettes, B: Non-surgcal treatment with air abrasion device and C: Non-surgcal treatment with titanium curettes + air abrasion device. Initial clinical periodontal parameters of all patients will be recorded and PIOS samples will be obtained. Following appropriate treatments for the determined group, clinical indices will be recorded and PIOS sampling will be repeated in the 3rd and 6th months. IL-10, IL-17, RANKL, OPG and TWEAK levels in the PIOS samples will be determined by ELISA test and the findings will be evaluated with appropriate statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Who have not received any periodontal treatment in the last 6 months,
2. Who have not used any medication (antibiotics, anti-inflammatory drugs, antibacterial mouthwashes, corticosteroids) that could affect the results of the study in the last 3 months,
3. Who have at least one implant with a probing depth of 6 mm or deeper in one or more areas in the mouth, and the implant in question has been in function for at least 1 year,
4. Between the ages of 18-65,
5. Individuals who approve the informed consent form will be included in the study.

Exclusion Criteria:

Individuals who:

1. have a systemic disease that may affect the periodontium,
2. regularly use medication that may affect the periodontium,
3. smoke,
4. are pregnant or lactating,
5. are sensitive to chlorhexidine,
6. have more than 50% bone loss around their current implant(s),
7. do not approve the informed consent form will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Probing Depth | From enrollment to the 6 months after treatment.
  The distance between the gingival margin and the base of the pocket will be measured with a periodontal probe.
Bleeding on probing | From enrollment to the 6 months after treatment
  Bleeding occurring within 10 seconds after probing will be evaluated as dichotomous (+/-).

SECONDARY OUTCOMES:
IL-10, RANKL, OPG, TWEAK, and IL-17 | 3rd and 6th months after treatment
  IL-10, RANKL, OPG, TWEAK, and IL-17 levels will be analyzed by ELISA test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided